CLINICAL TRIAL: NCT01297686
Title: A Clinical Trial of a Multi-Element Exercise Program for Plantar Fasciopathy in Workers Required to Stand for Prolonged Periods of Time
Brief Title: Exercise Versus Corticosteroid Randomized Clinical Trial for Plantar Fasciitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-03368; RS2010-IG20 (Other Grant/Funding Number: WorkSafeBC)
Record Dates: First submitted 2011-02-14; First posted 2011-02-17 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Fasciitis, Plantar
Keywords: Chronic plantar fasciitis; Workplace injury; Foot and Ankle Disability Index; Ultrasound measure of disease severity
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Multi-element exercise protocol involving static and dynamic stretches, deep massage, and balance training.
  Interventions: Other: Karaoke Exercise; Other: Balance walking exercise; Other: Forefoot extension exercise; Other: Standing one-legged balance exercise:; Other: Ankle inversion/eversion exercise; Other: Gastrocnemius and soleus stretching; Other: Tissue-specific plantar fascia self massage
- Standard of Care (Active Comparator): This arm will consist of a single injection of a corticosteroid, followed by stretching exercises for the calf.
  Interventions: Other: Gastrocnemius and soleus stretching; Drug: Dexamethasone

INTERVENTIONS:
Other: Karaoke Exercise — lateral side step movement involving crossing one foot over the next for 5 sets of 15 cross-overs in each direction
  Arms: Exercise
Other: Balance walking exercise — Walking along a straight line on the ground, for 5 sets of 30 strides
  Arms: Exercise
Other: Forefoot extension exercise — The subject stands feet shoulder width apart with one foot ahead of the other and then contracting only calf muscles of the back leg, lifts the heel of the back leg until the metatarsophalangeal joint of that foot is maximally extended. The subject is instructed to concentrate on maintaining balance on the back leg over the first and second metatarsophalangeal joints throughout movement for 5 sets of 15 repetitions.
  Arms: Exercise
Other: Standing one-legged balance exercise: — This exercise is performed initially with eyes open, then with mastery exhibited by being able to hold balance and not touch the ground with contralateral leg performed with eyes closed, then on an unstable surface with and without eyes open for 1 minute.
  Arms: Exercise
Other: Ankle inversion/eversion exercise — The foot is placed sideways at the edge of a step. After stabilizing the remainder of the foot and leg, the ankle is inverted and everted to the limits of the range for 3 sets of 15 repetitions.
  Arms: Exercise
Other: Gastrocnemius and soleus stretching — This stretch is performed while standing in a neutral position and the knee extended the foot is placed on top of a ramp or phone-book elevating the forefoot on the rearfoot (talocrural dorsiflexion) and held for 3 sets of 30 seconds each. Next the foot is again placed on top of a phone-book with the knee flexed approximately 15-20 degrees and held for 3 sets of 30 seconds each.
Other: Tissue-specific plantar fascia self massage — This deep massage is performed in a sitting position the right foot is crossed over the left while one hand passively extends the right forefoot. The left hand then applies light to moderate pressure in 3-5 second intervals along the length of the medial longitudinal arch. Same procedure is then repeated for the left foot.
  Arms: Exercise
Drug: Dexamethasone — A 22-gauge, 1.5" needle and 3 cm syringe filled with 1ml of dexamethasone mixed with 0.5ml of 1% lidocaine. Prior to injection, the skin will be sterilized with povidone-iodine. The needle is inserted 2-3 cm anteromedial to the focal point of pain in the inferior heel near the calcaneal tuberosity and moved toward the tenderest area.
  Arms: Standard of Care

SUMMARY:
Chronic plantar fasciopathy is a painful condition common in the workplace, particularly for those workers required to stand for long periods of time, and is typically associated with point tenderness at heel and arch of the foot. This clinical trial will investigate the effectiveness of an innovative multi-element exercise program versus the standard of care for plantar fasciopathy. The observation period will be 12-weeks. Outcomes are determined through questionnaire and ultrasound imaging. Workers with long-standing plantar fasciopathy who must stand for prolonged periods of time (i.e. > 6 hours) during their workday will be invited to participate in this study. After ensuring eligibility, each subject will be randomly assigned to either the intervention group who will receive a multi-element exercise program, or the control group who will receive a cortisone injection followed by a stretching program for their calf-muscles (standard of care). The treatment length for both groups will be 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult workers (men and women) between the ages of 19 and 60
* Workers required to stand for 6 hours or more in their respective workplaces
* Diagnosed with plantar fasciopathy (plantar fasciitis). All diagnoses will be made by a physiotherapist based on the presentation of palpable pain at or around the plantar medial heel, in addition to pain during weight-bearing activities and the presence of morning pain.
* Only individuals with pain for longer than 12 months will be included.

Exclusion Criteria:

* A history of surgery to their plantar fascia
* Osteoarthritis or other degenerative musculoskeletal disorders affecting the lower extremity
* Individuals who have received corticosteroid injections into their affected plantar fascia at any time in the past will be excluded.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Foot and Ankle Disability Index (FADI) at 6 weeks | 6 weeks
  Patient-centered health-realted quality of life indicator measuriing disability at the foot and ankle.
Change from Baseline in Foot and Ankle Disability Index (FADI) at 12 weeks | 12 weeks
  Patient-centered health-realted quality of life indicator measuriing disability at the foot and ankle.

SECONDARY OUTCOMES:
Change in Ultrasound-Based Grading of Pathology at 12 weeks | 12 weeks
  A 3-level ordinal scale assessing a composite of hypoechogenicity and neovascularity will be documented.
Change in Acoustoelastographic Analysis of Plantar Fascia Elasticity at 12 Weeks | 12 weeks
  A novel method of calculating the mechanical properties of deformation dependent soft-tissue using only ultrasound cine-images. Specific outcomes will include plantar fascial stiffness, strain, and modulus of elasticity.
Change in Visual Analog Scale for Pain at 12 weeks | 12 weeks
  Participants mark on a 100mm line the amount of pain on average they have experienced over the past 7 days. Items for both pain at work and pain with activities of daily living are included.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Taunton, Dr., Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada